CLINICAL TRIAL: NCT04665297
Title: An Individualized Approach to Promote Nurturing Care in Low and Middle Income Countries: A Hybrid Effectiveness/Implementation Trial of the International Guide for Monitoring Child Development
Brief Title: A Hybrid Effectiveness/Implementation Trial of the International Guide for Monitoring Child Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Mahatma Gandhi Institute of Medical Sciences (Other); Ummeed Child Development Center (Unknown); Ankara University (Other); Wuqu' Kawoq, Maya Health Alliance (Other); Harvard Medical School (HMS and HSDM) (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Peter J. Rohloff, M.D.,Ph.D., Assistant Professor/Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020P002143
Record Dates: First submitted 2020-12-02; First posted 2020-12-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Child Development
Keywords: Guatemala; India; Early Child Development

STUDY DESIGN:
Intervention Model Description: Nonblinded, two-arm cluster randomized controlled trial for 12 months. At 12 months, control arm crosses into the intervention, and both arms receive the intervention for an additional 12 months (total of 24 months)
Masking Description: Given nature of study, blinding is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Subjects from intervention clusters will receive the GMCD intervention, delivered in monthly visits to the home by frontline health workers, for 24 months. 0-12 months represents the primary effectiveness study, and 12-24 months a secondary maintenance study.
  Interventions: Behavioral: International Guide for Monitoring Child Development
- Control Arm (No Intervention): Subjects in control clusters will continue to receive usual care from their frontline health workers. After 12 months (primary effectiveness study) control will cross into the intervention for months 12-24.

INTERVENTIONS:
Behavioral: International Guide for Monitoring Child Development — Monthly GMCD visits includes assessment of risk factors, open-ended exploration of caregiver concerns about development, assessment of functioning in seven developmental domains, and using mutual problem solving strategies to develop a nurturing care plan with the caregiver.
  Arms: Intervention arm

SUMMARY:
The aim of this study is to conduct a hybrid effectiveness/implementation assessment of the International Guide for Monitoring Child Development (GMCD) in two LMIC settings, India and Guatemala, within established rural CHW programs. The primary objectives are (a) to evaluate the real-world effectiveness of the GMCD; (b) to use an implementation science framework to understand barriers and facilitators to effective population coverage, provider implementation, and maintenance; (c) to conduct an economic evaluation of the GMCD.

DETAILED DESCRIPTION:
Specific Aim 1: Assess the effectiveness of the GMCD intervention to improve developmental outcomes and nurturing care in India and Guatemala. The investigators will conduct a parallel-arm cluster randomized trial within rural CHW programs. In the primary effectiveness phase, children under 2 years old will receive the GMCD intervention or control for 12 months. Subsequently, control clusters will cross into the intervention, and continue an additional 12 months (total 24 study months). The primary developmental effectiveness outcome will be change in age-adjusted scores at 12 months on the Bayley Scales of Infant Development, 4th Edition BSID4) (3). The secondary nurturing care effectiveness outcome will be change in mean Home Observation for Measurement of the Environment (HOME) score at 12 months (4).

Specific Aim 2: Assess barriers and facilitators to GMCD implementation using the RE-AIM evaluation framework (5). RE-AIM domains will be assessed as: (a) Reach: participation rates, comparison of participant/non-participant characteristics, attendance/drop-out; (b) Effectiveness: impact on development (BSID4) and nurturing environment (HOME) [in Aim 1]; (c) Adoption: proportion of workers/facilities participating, CHW characteristics; (d) Implementation: contact hours/visit completion, fidelity to delivery protocols; (e) Maintenance: patient outcomes and cost effectiveness analysis at 12-24 months [in Aim 3]; intent by decision makers and implementers to continue intervention. In addition, the investigators will conduct a sequential quantitative-->qualitative explanatory analysis, using interviews and focus groups with implementers from clusters with highest/lowest impact outcomes (BSID4/HOME) to explore institutional inner and outer setting and implementation processes associated with intervention success, using the Consolidated Framework for Implementation Research (CFIR).

Specific Aim 3: Conduct an economic evaluation of the GMCD intervention. Evaluation will assess (a) costs of the interventions at 12 and 24 months; and (b) cost-effectiveness of the intervention (dollar per unit increase in BSID or HOME scores) at 12 months. This analysis will provide cost information to policymakers to help guide resource allocation decisions for ECD interventions.

ELIGIBILITY:
Inclusion Criteria:

* age 0-24 months at the time of enrollment visit
* receiving health services from frontline health workers of Maya Health Alliance (Guatemala), Mahatma Gandhi Institute (India) or their local partners

Exclusion Criteria:

* children who are critically ill and are judged by the frontline health worker to require hospitalization or center-based care
* children whose caregivers do not provide informed consent for the study

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 624 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Composite Language Score at 12 months | Change from 0 to 12 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 47-153
Change in Composite Motor Score at 12 months | Change from 0 to 12 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 46-154
Change in Composite Cognitive Score at 12 months | Change from 0 to 12 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 55-145

SECONDARY OUTCOMES:
Change in the Home Observation for Measurement of the Environment Scale (HOME) Raw Score | Change from 0 to 12 months
  Raw score range 0-45, higher scores better

OTHER OUTCOMES:
Change in Composite Language Score at 24 months | Change from 0 to 24 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 47-153
Change in Composite Motor Score at 24 months | Change from 0 to 24 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 46-154
Change in Composite Cognitive Score at 24 months | Change from 0 to 24 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 55-145
Change in the Home Observation for Measurement of the Environment Scale (HOME) Raw Score | Change from 0 to 24 months
  Raw score range 0-45, higher scores better

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rohloff, Principal Investigator — Assistant Professor/Associate Physician
Locations (2):
- Wuqu' Kawoq, Tecpán Guatemala, Guatemala
- Mahatma Gandhi Institute of Medical Sciences, Sevāgrām, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
We will deposit the above data in the Harvard Dataverse (https://dataverse.harvard.edu/) or another suitable public data repository, and it will be freely available there for any researcher wishing to perform secondary analysis, confirmation of primary study findings, or meta-analysis who adheres to the existing policy and procedures of the repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will submit data sets to the repository no later than 3 years after completion of final patient follow-up, or 2 years after the publication of the main study paper, whichever comes first.
Access Criteria: Publically available

REFERENCES:
- [Background] Ertem IO, Krishnamurthy V, Mulaudzi MC, Sguassero Y, Balta H, Gulumser O, Bilik B, Srinivasan R, Johnson B, Gan G, Calvocoressi L, Shabanova V, Forsyth BWC. Similarities and differences in child development from birth to age 3 years by sex and across four countries: a cross-sectional, observational study. Lancet Glob Health. 2018 Mar;6(3):e279-e291. doi: 10.1016/S2214-109X(18)30003-2. PMID 29433666
- [Background] Ertem IO, Dogan DG, Gok CG, Kizilates SU, Caliskan A, Atay G, Vatandas N, Karaaslan T, Baskan SG, Cicchetti DV. A guide for monitoring child development in low- and middle-income countries. Pediatrics. 2008 Mar;121(3):e581-9. doi: 10.1542/peds.2007-1771. PMID 18310178
- [Derived] Raut A, Mustafayev R, Srinivasan R, Chary A, Ertem I, Grazioso MDP, Gupta S, Krishnamurthy V, Lu C, Maliye C, Miller AC, Wagenaar BH, Rohloff P. Hybrid type 1 effectiveness/implementation trial of the international Guide for Monitoring Child Development: protocol for a cluster-randomised controlled trial. BMJ Paediatr Open. 2021 Sep 15;5(1):e001254. doi: 10.1136/bmjpo-2021-001254. eCollection 2021. PMID 34604546